CLINICAL TRIAL: NCT04438850
Title: Randomized, Double-blind, Multi Centre Phase II, Proof of Concept, Dose Finding Clinical Trial on Ivermectin for the Early Treatment of COVID-19
Brief Title: COVidIVERmectin: Ivermectin for Treatment of Covid-19
Acronym: COVER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Incidence has dramatically dropped and there is lack of eligible patients
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: cover_1
Record Dates: First submitted 2020-04-10; First posted 2020-06-19 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: ivermectin
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Ivermectin and placebo treatment will be double blinded, i.e. the treatment will be unknown to both the subject and the treating physician. The hospital pharmacist will be unblinded to study treatment because in charge to prepare the study treatment according to randomization arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- I_600 (Experimental): ivermectin 600 μg/kg daily for 5 consecutive days (I_600) + placebo
  Interventions: Drug: Ivermectin
- I_1200 (Experimental): ivermectin 1200 μg/kg daily at empty stomach with water for 5 consecutive days
  Interventions: Drug: Ivermectin
- Placebo (Placebo Comparator): placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ivermectin — Patients will be administered a single oral daily dose of approximately 600 μg/Kg (486-679 μg/Kg as rounded to a whole number of tablets), or 1200 μg/Kg (1098-1286 μg/Kg).
  Other Names: Ivermectin 9 mg cp by Chemo group
  Arms: I_1200; I_600
Other: Placebo — Patients should take placebo orally on an empty stomach with water
  Other Names: Placebo supplied by chemo group
  Arms: Placebo

SUMMARY:
Prospective, multi-centre, randomized, double-blind trial to assess efficacy and safety of ivermectin for the treatment of initial infection with SARS-CoV2 infection.

Study arms: A) placebo B) ivermectin 600 μg/kg daily for 5 consecutive days (I_600) + placebo. C) ivermectin 1200 μg/kg daily at empty stomach with water for 5 consecutive days (I_1200). Patients will be randomized at emergency room of hospitals as well as at outpatient ambulatory care as well as at home, according to routine procedures of recruiting centres.

In arm A and B, the number of placebo tablets to be administered will be calculated by the study dedicated pharmacist considering the number of tablets that should be taken in case a patient with the same weight is assigned to arm C.

DETAILED DESCRIPTION:
Primary objectives

The study is aimed:

1. at defining if ivermectin, administered at dosage of 600 μg/kg or 1200 μg/kg QD for five consecutive days is safe in patients with initial, asymptomatic or oligosymptomatic SARS_CoV-2 infection,
2. at defining if ivermectin, administered at the dosage(s) found to be safe decreases the viral load of SARS-CoV-2 at Day 7.

Secondary objectives To assess

1. the temporal profile of viral load at baseline, day 7, 14 and 30
2. the time to clinical cure (for symptomatic patients)
3. the proportion of patients with virological clearance at day 14 and 30.
4. the hospitalization rate.
5. the COVID-19 Severity Score at day 14 and 30

STUDY DESIGN

This is a multicentre, prospective, randomized, double-blind, adaptive phase II dose finding study.

Patients meeting the inclusion criteria will be asked to participate to the study and randomized in a 1:1:1 ratio to either:

* Placebo arm (arm A): placebo will be identical in appearance to ivermectin in order to preserve blinding and will be administered p.o. at empty stomach with water once daily, for 5 days
* Intervention arms: a) Ivermectin, single dose 600 μg/kg, for 5 days (I_600) and placebo (arm B) ; b) Ivermectin, single dose 1200 μg/kg, for 5 days (I_1200) (arm C) ); these drugs will be administered p.o. once daily, for 5 days.

In arm A and B, the number of placebo tablets to be administered will be calculated by the study dedicated pharmacist considering the number of tablets that should be taken in case a patient with the same weight is assigned to arm C.

Patients will be randomized by a centralized computer system. At randomization a treatment ID is assigned to the patient. Once a treatment ID is assigned this must not be re-assigned even in cases of errors.

Enrolled subjects will be identified by a unique subject number (patient code) that will remain consistent for the duration of the study.

Patients will be recruited at the emergency room of hospitals, and/or among asymptomatic hospital workers found positive for SARS-CoV-2 at routine screening and/or in outpatient ambulatory settings, and/or at home, if not meeting the clinical criteria for hospitalization, according to the routine procedure of each participating site. The expected duration of subject inclusion in the study is of 1 month, or until the planned number of subjects to be enrolled will be reached.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Positivity at RT-PCR per SARS_CoV2 (nasopharyngeal swabs)
* Consent to participation to the study and to the processing of personal data
* COVID-19 Severity Score < 3
* Patient able to take oral drugs

Exclusion Criteria:

* Pregnant or lactating women (pregnancy test not required, if doubt patient is excluded)
* Subjects suffering from known CNS diseases
* Lack of (or inability to provide) informed consent
* Patient under dialysis
* Any severe medical condition with a prognosis of < 6 months
* Patients under warfarin treatment
* Patients under antiviral treatment
* Patients under chloroquine phosphate or hydroxychloroquine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
SADR | 14 days
  Number of serious adverse drug reaction
Viral load | Assessed at day 7
  Quantitative viral load as measured by quantitative, digital droplet PCR.

SECONDARY OUTCOMES:
Trend viral load | Days 7 and 14 from baseline
  1. Trend over time of quantitative viral load at Day 7 and 14 as measured by quantitative, digital droplet PCR.
Clinical resolution | Assessed on Day 30
  Time to clinical resolution (for symptomatic patients).
Viral clearance | assessed on days 14 and 30
  Time from diagnosis to documented viral clearance
Virological clearance | Assessed at day 14 and 30
  Proportion of patients with virological clearance
hospitalization rate | Day 30
  rate of hospitalization
Severity score | Assessed at Day 14 and Day 30
  COVID-19 Severity Score (Coronavirus Diseases 19 Severity Score) - min value 1 ("no limitation of activities), max value 8 ("death"). Higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Zeno Bisoffi, Principal Investigator — IRCCS Sacro Cuore Don Calabria hospital
Locations (5):
- Italy (5):
  - IRCCS Sacro Cuore Don Calabria hospital, Negrar, Verona
  - Policlinico S. Orsola, Bologna
  - Ospedale Luigi Sacco, Milan
  - Ospedale di Rovereto, Rovereto
  - Ospedale Amedeo di Savoia, Turin

IPD SHARING:
Plan to Share IPD: Yes
The anonymized database will be uploaded into a public repository
Supporting Information: Study Protocol
Time Frame: The database will be available upon publication of the results
Access Criteria: The data will be available in a public repository